CLINICAL TRIAL: NCT00433212
Title: Efficacy and Safety of NIPPV to Increase Survival Without Bronchopulmonary Dysplasia in Extremely Low Birth Weight Infants
Brief Title: Nasal Intermittent Positive Pressure Ventilation in Premature Infants (NIPPV)
Acronym: NIPPV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NTG-2007-NIPPV; CIHR MCT-80246; ISRCTN15233270
Record Dates: First submitted 2007-02-07; First posted 2007-02-09 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Respiratory Insufficiency of Prematurity
Keywords: prematurity; respiratory insufficiency; non-invasive ventilation; bronchopulmonary dysplasia; hyaline membrane disease
MeSH Terms: conditions — Respiratory Insufficiency; Premature Birth; Bronchopulmonary Dysplasia; Hyaline Membrane Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Non-invasive respiratory support via nasal intermittent positive pressure ventilation
  Interventions: Device: NIPPV
- B (Active Comparator): Non-invasive respiratory support via nasal Continuous Positive Airway Pressure
  Interventions: Device: nCPAP

INTERVENTIONS:
Device: nCPAP — Deliver non-invasive respiratory support via ventilator with nCPAP device
  Arms: B
Device: NIPPV — Deliver non-invasive respiratory support via ventilator with NIPPV device
  Arms: A

SUMMARY:
The machines and oxygen used to help very premature babies breathe can have side-effects, such as bronchopulmonary dysplasia (BPD). Infants with BPD get more complications (a higher death rate, a longer time in intensive care and on assisted ventilation, more hospital readmissions in the first year of life, and more learning problems) than infants who do not develop BPD. Doctors try to remove the tube in the wind-pipe that links the baby to the breathing machine as soon as possible. However, small babies get tired, and still require help to breathe. One of the standard and common techniques to help them breathe without a tube in the wind-pipe is to use simple pressure support, nasal continuous positive airway pressure or nCPAP. This supports breathing a little, but it is often not enough to prevent the need to go back on the breathing machine.

Nasal intermittent positive pressure ventilation (NIPPV) is similar to nCPAP, but also gives some breaths, or extra support, to babies through a small tube in the nose. NIPPV is safe and effective, and already in use as an alternate "standard" therapy.

The main research question: After being weaned from the breathing machine, is NIPPV better than nCPAP in preventing BPD in premature babies weighing 999 grams or less at birth?

DETAILED DESCRIPTION:
The immature lung of extremely low birth weight (ELBW, < 1000 g) infants is easily damaged by the placement of an endotracheal tube to deliver mechanical ventilation and oxygen. This and the total time of mechanical ventilation contributes to bronchopulmonary dysplasia (BPD). Infants with BPD have an increased risk of later death or neuro-impairment. With the increasing survival of ELBW infants in the NICU, there has been a proportionate increase in the number of infants surviving with BPD.

Following invasive ventilation via an endotracheal tube (ETT), extubation to nasal Continuous Positive Airway Pressure (nCPAP)ventilation is the standard approach. Currently, 40% of infants who are extubated and given nCPAP support fail, and require re-intubation. Previous work suggests that a less invasive respiratory support such as Nasal Intermittent Positive Pressure Ventilation (NIPPV), without an endotracheal tube is less injurious to the lung. NIPPV may thereby reduce the duration of invasive ventilator support, and aid successful early extubation. We hypothesize that the use of NIPPV leads to a higher rate of survival without BPD than standard therapy with nCPAP.

This randomized clinical trial is appropriately powered to compare NIPPV with nCPAP to detect effects on clinically relevant long-term outcomes, such as death and BPD at 36 weeks. This is a multi-national, randomized, open clinical trial of two different standard methods of providing non-invasive respiratory support to 1000 extremely preterm infants weighing less than 1000 grams at birth.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight <1000 gm
* Gestational age <30 completed weeks
* Intention to manage the infant with non-invasive respiratory support (i.e. no endotracheal tube), where either:

  * the infant is within the first 7 days of life and has never been intubated or has received less than 24 hours of total cumulative intubated respiratory support;
  * the infant is within the first 28 days of life, has been managed with intubated respiratory support for 24 hours or more and is a candidate for extubation followed by non-invasive respiratory support.

Exclusion Criteria:

* Considered non-viable by clinician (decision not to administer effective therapies)
* Life-threatening congenital abnormalities including congenital heart disease (excluding patent ductus arteriosis)
* Infants known to require surgical treatment
* Abnormalities of the upper and lower airways
* Neuromuscular disorders
* Infants who are >28 days old and continue to require mechanical ventilation with an endotracheal tube

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1011 (Actual)
Dates: Start 2007-04; Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Composite of survival to 36 weeks gestational age, free of moderate-severe bronchopulmonary dysplasia | 36 weeks gestational age

SECONDARY OUTCOMES:
All cause mortality at 36 weeks gestational age | 36 weeks gestational age
All cause mortality before first discharge home | first discharge home
retinopathy of prematurity | discharge home
ultrasonographic evidence of brain injury | 36 weeks gestional age
necrotizing enterocolitis | 36 weeks gestational age
growth | discharge home
time to establish full feeds | discharge home
nosocomial infections | discharge home
need for re-intubation | 36 weeks gestational age
time on supplemental oxygen | discharge home
duration of positive pressure respiratory support | discharge home
comparison of synchronized and non-synchronized NIPPV | discharge home
bronchopulmonary dysplasia | 36 weeks gestational age
air leak syndromes | 36 weeks gestational age
nasal trauma | discharge home

CONTACTS AND LOCATIONS:
Overall Officials: Haresh Kirpalani, MD, MSc, Study Chair — Hamilton Health Sciences Corporation; Brigitte Lemyre, MD, Study Director — Children's Hospital of Eastern Ontario; Aaron Chiu, MD, Study Director — St. Boniface Hospital; David Millar, MD, Study Director — Royal Maternity Hospital, Belfast; Robin S Roberts, MTech, Study Director — Hamilton Health Sciences/McMaster University; Bradley Yoder, MD, Study Director — University of Utah; Peter H Dijk, MD, PhD, Study Director — University Medical Centrum Groningen
Locations (35):
- United States (14):
  - Georgetown University Children's Medical Center, Washington D.C., District of Columbia
  - The George Washington University Hospital, Washington D.C., District of Columbia
  - Tufts University Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center (BIDMC), Boston, Massachusetts
  - Virtua West Jersey Hospital, Voorhees Township, New Jersey
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Kings County Hospital, Brooklyn, New York
  - New York Hospital Queens, Brooklyn, New York
  - Queens Hospital Center, Jamaica, New York
  - Brookdale University Hospital & Medical Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Pennsylvania Hospital/U. of Pennsylvania, Philadelphia, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah
- LKH Feldkirch, Feldkirch, Austria
- CHC St. Vincent, Rocourt, Belgium
- Canada (8):
  - St. Boniface General Hospital/University of Manitoba, Winnipeg, Manitoba
  - Winnipeg Health Sciences Centre, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster University, Hamilton, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Ottawa Hospital General Campus, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Royal University Hospital, Saskatoon, Saskatchewan
- Ireland (3):
  - Cork University Maternity Hospital, Wilton, Cork
  - Coombe Women's Hospital, Dublin
  - National Maternity Hospital, Dublin
- Netherlands (2):
  - University Medical Center Groningen/Beatrix Children's Hosp, Groningen
  - Princess Amalia Dept of Pediatrics, Isala Clinics, Zwolle
- Hamad Medical Corporation, Doha, Qatar
- KK Women's and Children's Hospital, Singapore, Singapore
- Karolinska University Hospital/Astrid Lingrenn's Children's Hospital, Stockholm, Sweden
- United Kingdom (3):
  - Royal Maternity Hospital, Belfast, Northern Ireland
  - University of Leicester, Leicester
  - St. Mary's Hospital, London

REFERENCES:
- [Result] Kirpalani H, Millar D, Lemyre B, Yoder BA, Chiu A, Roberts RS; NIPPV Study Group. A trial comparing noninvasive ventilation strategies in preterm infants. N Engl J Med. 2013 Aug 15;369(7):611-20. doi: 10.1056/NEJMoa1214533. PMID 23944299
- [Derived] Bamat NA, Guevara JP, Bryan M, Roberts RS, Yoder BA, Lemyre B, Chiu A, Millar D, Kirpalani H. Variation in Positive End-Expiratory Pressure Levels for Mechanically Ventilated Extremely Low Birth Weight Infants. J Pediatr. 2018 Mar;194:28-33.e5. doi: 10.1016/j.jpeds.2017.10.065. Epub 2017 Dec 22. PMID 29275926
- [Derived] Millar D, Lemyre B, Kirpalani H, Chiu A, Yoder BA, Roberts RS. A comparison of bilevel and ventilator-delivered non-invasive respiratory support. Arch Dis Child Fetal Neonatal Ed. 2016 Jan;101(1):F21-5. doi: 10.1136/archdischild-2014-308123. Epub 2015 Jul 10. PMID 26162889